CLINICAL TRIAL: NCT00993057
Title: Comparing Two Glucose Sampling Frequencies for an Intensive Insulin Protocol During Craniotomy in Non-Diabetic Patients-How Efficiently and Safely Can We Maintain Target Glucose Levels
Brief Title: Efficiency of Two Glucose Sampling Protocols for Maintenance of Euglycemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Bebawy, Assistant Professor in Anesthesiology and Neurological Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00009023
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Brain Neoplasms; Intracranial Aneurysm
Keywords: Euglycemia; craniotomy; neurosurgery; hypoglycemia; insulin
MeSH Terms: conditions — Brain Neoplasms; Intracranial Aneurysm; Hypoglycemia; Insulin Resistance | interventions — Insulin; Insulin, Regular, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q1 hour protocol (Active Comparator): change of insulin infusion every hour
  Interventions: Drug: Insulin
- Q30min protocol (Active Comparator): change of insulin infusion every 30 minutes
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Adjustable insulin infusion scale with loading doses
  Other Names: Humulin

SUMMARY:
What is the efficacy and safety of q 30 minutes vs. q 1hour glucose sampling and intervention for an intensive insulin protocol to achieve and maintain euglycemia in non-diabetic patients undergoing craniotomy? The investigators hypothesize that in non-diabetic patients undergoing craniotomy, monitoring glucose and modifying insulin infusions every 30 minutes compared to every hour will help them reach target glucose levels faster and maintain them more efficiently with the same insulin protocol.

DETAILED DESCRIPTION:
Intraoperative blood glucose levels will be maintained in the target range of 90-110 mg/dL (euglycemia) using the protocol. The target serum glucose ranges chosen (90-110 mg/dL) was chosen to specifically target those levels associated with the best outcome in cerebral aneurysm surgery (serum glucose < 108 mg/dL) and aggressively avoid those levels associated with cognitive dysfunction (serum glucose < 128 mg/dL) and gross neurologic deficits (serum glucose < 152 mg/dL). Because the strength of these data, the investigators utilize an aggressive insulin protocol in their routine clinical care of patients undergoing craniotomies.

Each patient will be randomly assigned to one of two frequency of intervention groups-Group 30 will have the insulin dose adjusted every 30 minutes and Group 60 will have the insulin dose adjusted every 60 minutes. Blood glucose levels, insulin boluses and infusion rates, and dextrose boluses will be recorded on the respective Intraoperative Insulin & Glucose data sheet (Appendix 2 and 3 for Group 30 and Group 60, respectively).

Regardless of the protocol, glucose measurements will be conducted every 15 minutes but insulin intervention will be done at 30 minutes or one hour (per assigned treatment group). The interval data (15 minutes for the 30 min group and 15, 30, and 45 minutes for the 1 hour group) will be utilized to determine the pharmacodynamic effects of insulin (dose-response relationship). Interventions will only be performed at the assigned interval (30 vs 60 min) unless the glucose level is < 70 mg/dL, at which time the patient will receive 25 mL of 50% Dextrose solution. For these rescued patients, the protocol will be continued as scheduled.

On the day of surgery, after confirming entry into the study (i.e., confirmation of research consent), each patient will be randomly assigned to a specific protocol-q 30 minutes glucose measurements and intervention vs. q 60 minutes glucose measurements and intervention.Randomization will be performed in blocks of 10 using a computer generated random number assignment (odd numbers = q 30 minutes and even numbers = q 60 minutes)

ELIGIBILITY:
Inclusion Criteria:

* All English speaking, non-diabetic, non-pregnant patients over the age of 18 undergoing open craniotomy for the surgical treatment of tumors or intracranial aneurysms.

Exclusion Criteria:

* Patients under 18 years of age, patients who are pregnant, patients with diabetes, BMI > 33 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
performance of each of glucose sampling and insulin protocols for achieving euglycemia | duration of operation
  performance of each of glucose sampling and insulin protocols for achieving euglycemia during the operation

SECONDARY OUTCOMES:
hypoglycemia | duration of operation
  Hypoglycemia occurring the operation
time required to reach euglycemia | durarion of operation
  Elapsed time required to reach euglycemia during the operation
relationship of BMI and performance of protocols | duration of operation
  Evaluating the relationship of BMI (Body Mass Index) and the performance of protocols during the operation
relationship of serum biomarkers of insulin resistance and performance of protocols | duration of operation
  Evaluating the relationship of serum biomarkers of insulin resistance and performance of protocols during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Dhanesh Gupta, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Dhanesh Gupta, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fukuda S, Warner DS. Cerebral protection. Br J Anaesth. 2007 Jul;99(1):10-7. doi: 10.1093/bja/aem140. PMID 17573393
- [Background] Lukins MB, Manninen PH. Hyperglycemia in patients administered dexamethasone for craniotomy. Anesth Analg. 2005 Apr;100(4):1129-1133. doi: 10.1213/01.ANE.0000146943.45445.55. PMID 15781533
- [Background] Lindsberg PJ, Roine RO. Hyperglycemia in acute stroke. Stroke. 2004 Feb;35(2):363-4. doi: 10.1161/01.STR.0000115297.92132.84. No abstract available. PMID 14757880
- [Background] Pasternak JJ, McGregor DG, Schroeder DR, Lanier WL, Shi Q, Hindman BJ, Clarke WR, Torner JC, Weeks JB, Todd MM; IHAST Investigators. Hyperglycemia in patients undergoing cerebral aneurysm surgery: its association with long-term gross neurologic and neuropsychological function. Mayo Clin Proc. 2008 Apr;83(4):406-17. doi: 10.4065/83.4.406. PMID 18380986
- [Background] Carvalho G, Moore A, Qizilbash B, Lachapelle K, Schricker T. Maintenance of normoglycemia during cardiac surgery. Anesth Analg. 2004 Aug;99(2):319-24, table of contents. doi: 10.1213/01.ANE.0000121769.62638.EB. PMID 15271698
- [Background] Geroldi D, Falcone C, Emanuele E. Soluble receptor for advanced glycation end products: from disease marker to potential therapeutic target. Curr Med Chem. 2006;13(17):1971-8. doi: 10.2174/092986706777585013. PMID 16842191
- [Background] Meng YX, Ford ES, Li C, Quarshie A, Al-Mahmoud AM, Giles W, Gibbons GH, Strayhorn G. Association of C-reactive protein with surrogate measures of insulin resistance among nondiabetic US from National Health and Nutrition Examination Survey 1999-2002. Clin Chem. 2007 Dec;53(12):2152-9. doi: 10.1373/clinchem.2007.088930. Epub 2007 Oct 19. PMID 17951292
- [Background] Olufadi R, Byrne CD. Clinical and laboratory diagnosis of the metabolic syndrome. J Clin Pathol. 2008 Jun;61(6):697-706. doi: 10.1136/jcp.2007.048363. PMID 18505888
- [Background] Yamauchi T, Kamon J, Waki H, Terauchi Y, Kubota N, Hara K, Mori Y, Ide T, Murakami K, Tsuboyama-Kasaoka N, Ezaki O, Akanuma Y, Gavrilova O, Vinson C, Reitman ML, Kagechika H, Shudo K, Yoda M, Nakano Y, Tobe K, Nagai R, Kimura S, Tomita M, Froguel P, Kadowaki T. The fat-derived hormone adiponectin reverses insulin resistance associated with both lipoatrophy and obesity. Nat Med. 2001 Aug;7(8):941-6. doi: 10.1038/90984. PMID 11479627
- [Background] Yudkin JS, Stehouwer CD, Emeis JJ, Coppack SW. C-reactive protein in healthy subjects: associations with obesity, insulin resistance, and endothelial dysfunction: a potential role for cytokines originating from adipose tissue? Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):972-8. doi: 10.1161/01.atv.19.4.972. PMID 10195925
- [Background] Varvel JR, Donoho DL, Shafer SL. Measuring the predictive performance of computer-controlled infusion pumps. J Pharmacokinet Biopharm. 1992 Feb;20(1):63-94. doi: 10.1007/BF01143186. PMID 1588504